CLINICAL TRIAL: NCT03369288
Title: Assessing Cement-bone Incorporation and Adjacent Segment Degeneration Following Cement Augmentation; an MRI-PET Follow-up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01207
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Vertebral Fracture; Cement Augmentation
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Intervention Model Description: Prospective PET-MRI follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET MRI — 18F-fluoride PET-MRI

SUMMARY:
3-year PET-MRI follow-up after vertebral balloon kyphoplasty aiming to investigate cement incorporation.

ELIGIBILITY:
Inclusion criteria

* Men and women aged 18 to 70 years
* Minimum 3-year follow-up
* Single-level vertebral kyphoplasty
* Index surgery at UniversitätsSpital Zürich
* MRI-scan during initial treatment
* Informed consent provided

Exclusion criteria

* Combined with other operative procedure on the spine (e.g. dorsal instrumentation)
* Intraoperative intradiscal cement leakage
* Previous history of spinal surgery except on the cervical spine
* Metastatic disease with skeletal involvement
* Known chronic diseases of the bone metabolism other than osteoporosis
* Documented pregnancy (see also 6.3)
* Presence of implants not suited for MRI (pacemaker, neuro-stimulators, pain pumps, insulin pumps, Cochlea implants, metallic foreign bodies like bullet fragments)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-06-28 (Estimated); Study Completion 2019-11-28 (Estimated)

PRIMARY OUTCOMES:
Tracer Uptake | at least 3 years after kyphoplasty
  Perifokal tracer uptake at the cement-bone border

SECONDARY OUTCOMES:
Intravertebral Discs | at least 3 years after kyphoplasty
  Tracer uptake within the intravertebral disc and morphological changes

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Trauma Surgery, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No